CLINICAL TRIAL: NCT06321939
Title: Sequencing-based Counting of Plasma Epstein-Barr Virus DNA in Non-metastatic Nasopharyngeal Carcinoma
Status: Recruiting | Type: Observational
Sponsor: Hunan Cancer Hospital (Other)
Responsible Party: Principal Investigator, Yaqian Han, Professor, Hunan Cancer Hospital
Other Study IDs: NPCNS 001
Record Dates: First submitted 2024-02-24; First posted 2024-03-20 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Nasopharyngeal Carcinoma; Herpesvirus 4, Human
MeSH Terms: conditions — Nasopharyngeal Carcinoma; Epstein-Barr Virus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: EBV-DNA next generation sequencing — EBV-DNA next generation sequencing

SUMMARY:
The investigators aim to explore a new EBV DNA surveillance method with both high sensitivity and specificity in nasopharyngeal carcinoma (NPC) patients. the investigators aim to conduct plasma EBV DNA counting by next generation sequencing (NGS) in non-metastatic NPC patients on their diagnose, after two cycles of induction chemotherapy (IC), and 4-8 weeks after definitive radiotherapy. The investigators aim to explore whether sequencing-based counting is better than PCR analysis in plasma EBV-DNA surveillance, so as to monitoring tumor responses to treatment and for guiding individualized treatment adaptation in the future.

DETAILED DESCRIPTION:
The investigators aim to explore a new EBV DNA surveillance method with both high sensitivity and specificity in nasopharyngeal carcinoma (NPC) patients. the investigators aim to conduct plasma EBV DNA counting by next generation sequencing (NGS) in non-metastatic NPC patients on their diagnose, after two cycles of induction chemotherapy (IC), and 4-8 weeks after definitive radiotherapy. The investigators aim to explore whether sequencing-based counting is better than PCR analysis in plasma EBV-DNA surveillance, so as to monitoring tumor responses to treatment and for guiding individualized treatment adaptation in the future.

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed, pathologically proven World Health Organization (WHO) type II/III untreated NPC;
2. Non-metastatic NPC (I-IVA, according to the 8th edition of the AJCC/UICC clinical staging system);
3. Age at diagnosis: over 18 years old;
4. Eastern Cooperative Oncology Group (ECOG) score: 0-1
5. Receiving recommended curative intention treatments：definitive radiotherapy w/wo three cycles of induction chemotherapy (IC) (gemcitabine-cisplatin [GP] or paclitaxel-cisplatin [TP] regimen);
6. Pre-treatment and post-IC1 cell-free Epstein-Barr virus (cfEBV) DNA > 0 copy/mL; systemic cfEBV DNA monitoring during IC phase for risk stratification;
7. Normal hematic, liver, and kidney function: hemoglobin (HG) > 90 g/L; neutrophil > 1.5 × 109/L; platelet > 100 × 109/L; total bilirubin (TBIL) ≤ 1.5 × upper limit of normal (ULN); alanine transaminase (ALT) and aspartate transaminase (AST) ≤ 2.5 × ULN; alkaline phosphatase (ALP) ≤ 2.5 × ULN; creatinine clearance (Ccr) ≥ 60 mL/min;
8. Female subjects capable of becoming pregnant agree to use reliable contraceptive measures from screening to 1 year after treatment;
9. Patients will be required to sign informed consent forms and be willing and able to comply with the requirements for visits, treatment, laboratory tests, and other research requirements stipulated in the research schedule.

Exclusion Criteria:

1. Receiving surgery, target therapy, and/or immunotherapy during or before induction phase;
2. Other previous or concurrent malignant tumors, except adequately treated non-melanoma skin cancer, cervical carcinoma in situ, and thyroid papillary cancer;
3. Pregnant or lactating women (a pregnancy test should be considered for fertile women with an active sex life);
4. Previously treated with radical radiotherapy (RT), except non-melanoma skin cancers outside intended RT treatment volume;
5. Uncontrolled heart disease, e.g.: 1) Heart failure, New York Heart Association (NYHA) level ≥ 2; 2) unstable angina; 3) myocardial infarction in the past 1 year; 4) supraventricular or ventricular arrhythmia requiring treatment or intervention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Non-metastatic NPC
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-01-11 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Positivity rate of plasma EpsteineBarr virus (EBV) DNA by next generation sequencing | from diagnose to 4-8 weeks after definitive radiotherapy
  Plasma EBV DNA analysis by NGS on enrollment, after 2 cycles of induction chemotherapy, and 4-8 weeks after definitive radiotherapy.

SECONDARY OUTCOMES:
Overall survival | 2 year
  Measured from the day of enrollment until death due to any cause, or the last follow-upmeasured from the day of enrollment until death due to any cause, or the last follow-up visit.
Distant metastasis failure-free survival | 2 year
  Measured from the day of enrollment until death until distant metastasis , or the last follow-up visit.
Locoregional failure-free survival | 2 year
  Measured from the day of enrollment until death until local and/or regional recurrence, or the last follow-up visit.
Failure-free survival | 2 year
  Measured from the day of enrollment until treatment failure, death from any cause, or the last follow-up visit, whichever occurred first.
Patient reported quality-of-life score | up to 2 years
  Patient reported quality of life would be evaluated using the Quality of Life Questionnaire-Core 30 module (QLQ-C30).
Biomarker analysis | from diagnose to 4-8 weeks after definitive radiotherapy
  Exploratory biomarker analysis that would be able to predict patient treatment benefits, for example PD-L1 expression, antigen (other than EBV, eg. human cytomegalovirus(human cytomegalovirus [HCMV], TTV) DNA counting.

CONTACTS AND LOCATIONS:
Locations (1):
- Hunan cancer Hospital, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No